CLINICAL TRIAL: NCT02121431
Title: Online vs Staff Delivery: Child & Family Outcomes, Value Analysis, Satisfaction
Brief Title: Child and Family Outcomes and Consumer Satisfaction for Online vs Staff-Delivered Parenting Intervention
Acronym: TPAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Carolina (Other)
Collaborators: Oregon Research Institute (Other); University of Georgia (Other); The University of Queensland (Other)
Responsible Party: Principal Investigator, Ron Prinz, PhD, Carolina Distinguished Professor, University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pro00024933
Record Dates: First submitted 2014-04-21; First posted 2014-04-23 (Estimated); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: Childhood Disruptive Behavior Disorders; Oppositional Defiant Disorder; Conduct Disorder; Attention Deficit Hyperactivity Disorder; Parent-Child Interactions
MeSH Terms: conditions — Oppositional Defiant Disorder; Conduct Disorder; Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Online-Delivered Parenting Intervention (Experimental): The Online-Delivered Parenting Intervention, which is based on the Triple P--Positive Parenting Program system of interventions, is an interactive website designed to engage and activate the participant through sequenced, personalized, interactive, and video-based content. The intervention emphasizes a self-regulatory process, parent specification of goals, practical and straightforward parenting strategies, modeling, and action activation.
  Interventions: Behavioral: Triple P--Positive Parenting Program
- Staff-Delivered Parenting Intervention (Active Comparator): The Staff-Delivered Parenting Intervention is based on the Triple P--Positive Parenting Program system and involves 10 face-to-face sessions with each family. This intervention is the well-established Level 4 Standard Triple P program.
  Interventions: Behavioral: Triple P--Positive Parenting Program

INTERVENTIONS:
Behavioral: Triple P--Positive Parenting Program — The Triple P--Positive Parenting Program (Triple P), which has an extensive evidence base, is grounded in a common set of core principles of positive parenting and draws on a broad menu of parenting strategies. A key provision of Triple P is that parents are the decision-makers about program goals and selection/implementation of specific parenting strategies consistent with their preferences and values.

SUMMARY:
This trial addresses a serious and all-too-frequent public health problem, namely early-onset disruptive behavior problems in young children. The focus is on testing an online treatment program which empowers parents to help their children to improve their mental health and behavioral functioning. At the conclusion of the study, the investigators will know whether the online-delivered program works as well as an established staff-delivered program, with respect to child disruptive behavior problems, parenting, parent/family stress, consumer satisfaction, and value analysis.

DETAILED DESCRIPTION:
High-prevalence mental health problems require innovative strategies to broaden reach of evidence-based services. Disruptive behavior problems (DBPs), or conduct problems, in young children represent a major public health challenge that is not only highly prevalent but also, left untreated, heighten risk for adverse mental health and developmental outcomes in adolescence and adulthood. Internet and online technology has considerable potential to help achieve such a goal. Building on parenting interventions that have demonstrated impact on childhood DBPs, this clinical trial compares an online-delivered intervention to a well-validated staff-delivered intervention, holding program content constant. Both interventions are based on the Triple P-Positive Parenting Program. The sample includes families with a 3-7 year old child who has a pronounced level of DBPs. The study makes use of a non-inferiority trial design to determine whether the online-delivered intervention yields as good outcomes as the well-established staff-delivered intervention with respect to childhood DBPs, parenting, and parent/family stress. The study also includes a value analysis comparing the two interventions, accounting for provider and participant expenses as well as pre-implementation and implementation phases. This study is intended to shed light on the impact and potential benefits of a viable online parenting intervention for childhood disruptive behavior problems, but the results from this study are also intended to help the mental health field to better understand more broadly the potential advantages and disadvantages of online interventions over traditionally delivered interventions, particularly in light of expense minimization/effectiveness analysis.

ELIGIBILITY:
Inclusion Criteria:

* clinically elevated level of child disruptive behavior problems
* parent resides with the child and has primary custody
* parent has access to internet via computer, e-tablet, or smartphone

Exclusion Criteria:

* already in a family-based treatment
* child has pervasive developmental disorder
* parent under 20 years of age
* parent has serious mental illness

Ages: 3 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 334 (Actual)
Dates: Start 2014-04; Primary Completion 2019-04-01 (Actual); Study Completion 2019-04-01 (Actual)

PRIMARY OUTCOMES:
childhood disruptive behavior problems | up to 12 months
  parental report; independent observation; teacher report

SECONDARY OUTCOMES:
parenting behavior | baseline, 4 months (T2), 12 months (T3)
  parental report; independent observation
parent and family stress | baseline, 4 months (T2), 12 months (T3)
  parenting daily hassles; impact on family quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Ronald J Prinz, Ph.D., Principal Investigator — University of South Carolina
Locations (2):
- United States (2):
  - Oregon Research Institute, Eugene, Oregon
  - Parenting & Family Research Center, University of South Carolina, Columbia, South Carolina

REFERENCES:
- [Derived] Ingels JB, Corso PS, Prinz RJ, Metzler CW, Sanders MR. Online-Delivered Over Staff-Delivered Parenting Intervention for Young Children With Disruptive Behavior Problems: Cost-Minimization Analysis. JMIR Pediatr Parent. 2022 Mar 11;5(1):e30795. doi: 10.2196/30795. PMID 35275084
- [Derived] Prinz RJ, Metzler CW, Sanders MR, Rusby JC, Cai C. Online-delivered parenting intervention for young children with disruptive behavior problems: a noninferiority trial focused on child and parent outcomes. J Child Psychol Psychiatry. 2022 Feb;63(2):199-209. doi: 10.1111/jcpp.13426. Epub 2021 Apr 8. PMID 33829499